CLINICAL TRIAL: NCT03346876
Title: Autonomic Dysfunction in Patients With Pectus Excavatum.
Acronym: ADPE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 05-XD-57-110; TCRD-TPE-106-RT-2 (Other Grant/Funding Number: Taipei Tzu-Chi Hospital, Buddhist Tzu-Chi Medical Foundation)
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-08

CONDITIONS: Pectus Excavatum; Autonomic Dysfunction; Surgery
Keywords: Pectus excavatum, heart rate variability
MeSH Terms: conditions — Funnel Chest; Primary Dysautonomias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: patients with pectus excavatum
  Interventions: Procedure: Nuss surgery
- Control group: healthy subjects without pectus excavatum

INTERVENTIONS:
Procedure: Nuss surgery — surgical correction for pectus excacatum
  Groups: Study group

SUMMARY:
Investigators conducted a pilot study to to evaluate the autonomic function in participants with pectus excavatum before and after Nuss surgery.

DETAILED DESCRIPTION:
Since pectus excavatum can cause cardiac arrhythmia, the cardiac autonomic function in participants with pectus excavatum might be impaired. However, to our knowledge, there is no any study to evaluate the cardiac autonomic function in participants with pectus excavatum.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of pectus excavatum
2. Agree to receive Nuss surgery to correct pectus excavatum

Exclusion criteria:

1. Major medical disease (asthma, heart failure, renal disease)
2. Known psychiatric disease
3. Known sleep-disordered breathing
4. Skeletal disease
5. Major surgery within 6 months

Ages: 13 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 13~45 y/o pectus patients and healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-07-31 (Estimated); Study Completion 2018-07-31 (Estimated)

PRIMARY OUTCOMES:
The impact of Nuss surgery on HRV in patients with pectus excavatum | 6 months
  If Nuss surgery can improve HRV in different stress in patients with pectus excavatum?

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Chen Yang, MD, Study Chair — Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Locations (1):
- Taipei Tzu-Chi Hospital, Buddhist Tzu-Chi Medical Foundation, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Tobaldini E, Nobili L, Strada S, Casali KR, Braghiroli A, Montano N. Heart rate variability in normal and pathological sleep. Front Physiol. 2013 Oct 16;4:294. doi: 10.3389/fphys.2013.00294. PMID 24137133
- [Derived] Hsu YT, Cheng YL, Chang YW, Lan CC, Wu YK, Yang MC. Autonomic nervous system dysregulation in response to postural change in patients with pectus excavatum in Taiwan: a pilot study. J Cardiothorac Surg. 2022 May 3;17(1):89. doi: 10.1186/s13019-022-01835-5. PMID 35505418